CLINICAL TRIAL: NCT06036108
Title: A Multicenter, Randomized, Open-label, 2-arm, 2-period Crossover Trial to Investigate the Effects of Food on the Pharmacokinetics of a Single Dose of Brexpiprazole Once-weekly (QW) Formulation in Patients With Schizophrenia
Brief Title: Food Effect Study of Brexpiprazole Once-weekly (QW) Formulation in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 331-102-00151
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting-state administration group (Experimental): Brexpiprazole QW formulation in a fasting-state administration
  Interventions: Drug: OPC-34712FUM/ Brexpiprazole fumarate
- Fed-state administration group (Experimental): Brexpiprazole QW formulation in a fed-state administration
  Interventions: Drug: OPC-34712FUM/ Brexpiprazole fumarate

INTERVENTIONS:
Drug: OPC-34712FUM/ Brexpiprazole fumarate — In Period 1, a single oral dose of two 24 mg tablets of brexpiprazole QW formulation (48 mg as brexpiprazole) will be administered at least 10 hours of fasting. In Period 2, following at least 10 hours of fasting, the subject will consume a high-fat meal within 20 minutes, after which a single oral dose of two 24 mg tablets of brexpiprazole QW formulation (48 mg as brexpiprazole) will be administered within 10 minutes of finishing the meal.
  Arms: Fasting-state administration group
Drug: OPC-34712FUM/ Brexpiprazole fumarate — In Period 1, following at least 10 hours of fasting, the subject will consume a high-fat meal within 20 minutes, after which a single oral dose of two 24 mg tablets of brexpiprazole QW formulation (48 mg as brexpiprazole) will be administered within 10 minutes of finishing the meal. In Period 2, a single oral dose of two 24 mg tablets of brexpiprazole QW formulation (48 mg as brexpiprazole) will be administered following at least 10 hours of fasting.
  Arms: Fed-state administration group

SUMMARY:
To investigate the effect of food on the pharmacokinetics of a single dose of brexpiprazole QW formulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia based on DSM-5® at the time of informed consent
* Patients who are able to be hospitalized for the protocol-defined hospitalization period
* Patients with a body mass index [BMI = body weight (kg)/height (m)²] of 18.5 kg/m² or higher and lower than 35.0 kg/m² at screening
* Patients who, in the judgment of the investigator, have stable psychotic symptoms maintained by administration of an antipsychotic within the dosing range indicated below, before commencement of IMP administration [Upper limit of dose and regimen] Antipsychotic medication comprising no more than 2 active components, and a daily dose equivalent to ≤600 mg/day of chlorpromazine
* Patients who are able to finish the high-fat meal specified in this protocol within 20 minutes

Exclusion Criteria:

* Patients with a concurrent mental disorder besides schizophrenia who are judged by the investigator to be unsuitable for participation in the trial
* Patients who have met the DSM-5® diagnostic criteria for substance-related or addictive disorder, including alcohol and benzodiazepines but excluding caffeine and tobacco, within 180 days before commencement of investigational medicinal product (IMP) administration
* Patients who fall under any of the following criteria regarding suicidal ideation and suicidal behavior

  * Patients who answered "yes" to Question 4 "Active Suicidal Ideation with Some Intent to Act, without Specific Plan" or Question 5 "Active Suicidal Ideation with Specific Plan and Intent" regarding C-SSRS suicidal ideation at screening (for the past 6 months) or at the Period 1 baseline examination (since the last assessment)
  * Patients who exhibited suicidal behavior on C-SSRS at screening (for the past 2 years) or at the Period 1 baseline examination (since the last assessment)
  * Patients who present a serious risk of suicide based on the judgment of the investigator
* Patients who have previously undergone gastrointestinal surgery that could affect PK evaluation
* Patients who have a clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorder. Medical conditions that are minor or well-controlled may be considered acceptable if the condition does not interfere with safety and PK assessments.
* Patients who are using clozapine at the time of informed consent
* Patients whose clinical symptoms have worsened to the point where use of prohibited concomitant therapy or medication is required during the washout period for prior medication
* Patients whose cytochrome P450 2D6 (CYP2D6) phenotype is judged to be either poor metabolizers (PM) or Unknown based on the results of CYP2D6 genotyping at screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Rainbow & Sea Hospital, Saga, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 59 participants from 26 trial sites in 1 countries.
Pre-assignment Details: Adults with schizophrenia as defined by Diagnostic and Statistical Manual of Mental Health Disorders 5th Edition Text Revision criteria were included.
Groups:
- Fasting-state Administration Preceding Group: Brexpiprazole QW formulatio in a fasting-state preceding administration
- Fed-state Administration Preceding Group: Brexpiprazole QW formulatio in a fed-state preceding administration
Period: Overall Study
Arm/Group | Fasting-state Administration Preceding Group | Fed-state Administration Preceding Group
Started | 29 | 30
Completed | 22 | 23
Not Completed | 7 | 7
Not completed — Adverse Event | 4 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Meets Study-Specific Discontinuation Criteria | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set, which included all randomized patients who received the study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasting-state Administration Preceding Group | Fed-state Administration Preceding Group | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 30 | 59
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.5 (10.9) | 49.8 (12.5) | 48.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 24 | 19 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 29 | 30 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Brexpiprazole in Plasma After Administration in a Fed State Versus Administration in a Fasting State
Description: To evaluate Cmax of brexpiprazole following single oral administration of brexpiprazole QW formulation in a fed state versus administration in a fasting state
Time Frame: PK: Pre-dose, 3, 9, 24, 36, 48, 72, 120, 168, 240, 312 hours post-dose
Population: The food effect analysis set includes all subjects for whom Cmax, AUC∞ or AUCt could be calculated throughout Period 1 and Period 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fasting-state Administration: Brexpiprazole QW formulatio in a fasting-state administration
- Fed-state Administration: Brexpiprazole QW formulatio in a fed-state administration
Arm/Group | Fasting-state Administration | Fed-state Administration
Number analyzed (Participants) | 45 | 45
ng/mL | 221.9 (108.2) | 365.2 (156.2)

2. Primary Outcome: Area Under Curve (AUC) of Brexpiprazole in Plasma After Administration in a Fed State Versus Administration in a Fasting State
Description: To evaluate AUC of brexpiprazole following single oral administration of brexpiprazole QW formulation in a fed state versus administration in a fasting state
Time Frame: PK: Pre-dose, 3, 9, 24, 36, 48, 72, 120, 168, 240, 312 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h∙ng/mL
Arm/Group | Fasting-state Administration | Fed-state Administration
Number analyzed (Participants) | 45 | 45
h∙ng/mL
  AUC infinity | 25400 (16200) | 37100 (20800)
  AUCt | 23400 (14100) | 34700 (18600)

ADVERSE EVENTS:
Time Frame: Adverse event are collected after a subject signs the ICF, and continue until the follow-up period, up to 112 days.
Description: An AE is defined as any untoward medical occurrence in a clinical trial subject administered a drug used in the clinical trial and which does not necessarily have a causal relationship with this treatment. In this trial, any untoward medical occurrence in a subject not administered a drug used in the clinical trial is also deemed as an AE.
Groups:
- Fasted Stated: Brexpiprazole QW formulatio in a fasting-state administration
- Fed Stated: Brexpiprazole QW formulatio in a fed-state administration
Arm/Group | Fasted Stated | Fed Stated
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/52 | 1/55
Other Adverse Events (participants affected / at risk) | 15/52 | 24/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fasted Stated (N=52) | Fed Stated (N=55)
Dystonia (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fasted Stated (N=52) | Fed Stated (N=55)
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 5 | 7
Vomiting (Gastrointestinal disorders) | 2 | 11
Malaise (General disorders) | 1 | 3
Nasopharyngitis (Infections and infestations) | 3 | 0
Dizziness (Nervous system disorders) | 1 | 5
Somnolence (Nervous system disorders) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT06036108/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT06036108/SAP_001.pdf